CLINICAL TRIAL: NCT01361295
Title: The Occurrence of Cerebral Embolism (CE) in Catheter Ablation of Atrial Fibrillation (AF) Using Two Different Ablation Catheters
Brief Title: Cerebral Embolism (CE) in Catheter Ablation of Atrial Fibrillation (AF)
Acronym: CE-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Serge A. Trines (Other)
Responsible Party: Sponsor-Investigator, Serge A. Trines, Senior cardiologist, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE-AF-002
Record Dates: First submitted 2011-05-20; First posted 2011-05-26 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; cerebral embolism; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation; Intracranial Embolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PVI with PVAC gold (Active Comparator): Patient for pulmonal vein isolation using the PVAC Gold Catheter. Intervention.
  Interventions: Procedure: PVI with Cooled-RF
- PVI with Cooled-RF (Active Comparator): Patient for pulmonal vein isolation using the Cooled-RF catheter.
  Interventions: Procedure: PVI with PVAC gold

INTERVENTIONS:
Procedure: PVI with PVAC gold — Pulmonary vein isolation using the Medtronic PVAC gold catheter
  Other Names: Medtronic AF solutions
  Arms: PVI with Cooled-RF
Procedure: PVI with Cooled-RF — Pulmonary vein isolation using the Biosense Webster Navistar Thermocool catheter
  Other Names: CARTO3 system
  Arms: PVI with PVAC gold

SUMMARY:
Radiofrequency catheter ablation of atrial fibrillation (AF) induces a procoagulant state, which leads to an acute risk for symptomatic cerebral embolism (CE) of approximately 1%. The induction of a procoagulant state has been studied in pulmonary vein isolation (PVI) with a non-cooled tip catheter. The induction of a procoagulant state using a cooled-tip catheter has not been studied yet. Due to the avoidance of high endocardial temperatures, it can be expected that these procedures induce a lower level of procoagulation.

Recent studies showed an 11% incidence of CE on diffusion weighted (DW) MRI in patients undergoing cooled-tip catheter ablation of AF. In this study there will be used to different catheters, the cooled-tip catheter and the PVAC Gold catheter. Since the PVAC Gold catheter is equipped with non-cooled electrodes, the risk of endothelial scarring, local thrombosis and CE may be increased.

The goal of this study is to determine the effect of two different ablation catheters on the induction of a procoagulant state and the incidence of CE on DW-MRI in patients with AF undergoing PVI.

Our hypothesis is that patients with AF undergoing PVI using the PVAC gold catheter will show a higher rise in procoagulation and a higher incidence of CE on DW-MRI than patients with AF undergoing PVI with the cooled-tip catheter.

DETAILED DESCRIPTION:
A total of 70 patients scheduled for a first ablation of paroxysmal AF will be included. Patients will be 1:1 randomized to PVI using the PVAC gold catheter or the cooled-tip catheter. A control group of 20 patients with AF but without undergoing ablation is included for neuropsychological testing.

Before the procedure, the procoagulant state will be assessed by measuring several markers of endothelial damage, activated coagulation, fibrinolysis and by measurement of fibrinogen and thrombin generation. Measurements will be repeated during and after the procedure.

Documentation of the formation of CE will be established by performing a DW-MRI before and after the ablation. The proportion of symptomatic CE will be quantified by neuropsychological tests and questionnaires.

Finally, transcranial doppler will be performed during the entire procedure to quantify the number and pattern of cerebral microembolic signals (MES).

ELIGIBILITY:
Inclusion Criteria:

* suffering from drug-refractory paroxysmal atrial fibrillation
* scheduled for first ablation procedure

Exclusion Criteria:

* contra-indications for DW-MRI
* previous AF-ablation
* minors
* any patient unable to undergo neuropsychological testing due to mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cerebral embolism | Between 24 hours before the ablation and 24 hours after the ablation
  Cerebral embolism will be documented with diffusion weighted MRI of the brain before and after ablation.

SECONDARY OUTCOMES:
Neuropsychological functioning | Between a week before the ablation until 3 months after the ablation
  A decrease in neuropsychological functioning will be assessed with a questionnaire before and after the procedure
Rise in procoagulation | Between 24 hours before the ablation and 24 hours after the ablation
  The procoagulant state will be assessed before, during and after the procedure by measurement of markers of endothelial damage, markers of activated coagulation, markers of fibrinolysis and by measurement of APTT, PT-INR, fibrinogen and thrombin generation.

CONTACTS AND LOCATIONS:
Overall Officials: Serge A. Trines, MD, PhD, Principal Investigator — Cardiology, LUMC
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

REFERENCES:
- [Background] Sauren LD, VAN Belle Y, DE Roy L, Pison L, LA Meir M, VAN DER Veen FH, Crijns HJ, Jordaens L, Mess WH, Maessen JG. Transcranial measurement of cerebral microembolic signals during endocardial pulmonary vein isolation: comparison of three different ablation techniques. J Cardiovasc Electrophysiol. 2009 Oct;20(10):1102-7. doi: 10.1111/j.1540-8167.2009.01509.x. Epub 2009 Jun 22. PMID 19549035
- [Background] Schrickel JW, Lickfett L, Lewalter T, Mittman-Braun E, Selbach S, Strach K, Nahle CP, Schwab JO, Linhart M, Andrie R, Nickenig G, Sommer T. Incidence and predictors of silent cerebral embolism during pulmonary vein catheter ablation for atrial fibrillation. Europace. 2010 Jan;12(1):52-7. doi: 10.1093/europace/eup350. PMID 19933517
- [Background] Bulava A, Slavik L, Fiala M, Heinc P, Skvarilova M, Lukl J, Krcova V, Indrak K. Endothelial damage and activation of the hemostatic system during radiofrequency catheter isolation of pulmonary veins. J Interv Card Electrophysiol. 2004 Jun;10(3):271-9. doi: 10.1023/B:JICE.0000026924.96281.be. PMID 15133367
- [Derived] Kece F, Bruggemans EF, de Riva M, Alizadeh Dehnavi R, Wijnmaalen AP, Meulman TJ, Brugman JA, Rooijmans AM, van Buchem MA, Middelkoop HA, Eikenboom J, Schalij MJ, Zeppenfeld K, Trines SA. Incidence and Clinical Significance of Cerebral Embolism During Atrial Fibrillation Ablation With Duty-Cycled Phased-Radiofrequency Versus Cooled-Radiofrequency: A Randomized Controlled Trial. JACC Clin Electrophysiol. 2019 Mar;5(3):318-326. doi: 10.1016/j.jacep.2018.11.008. Epub 2018 Dec 26. PMID 30898234